CLINICAL TRIAL: NCT04208607
Title: Bronchiectasis Phenotypes ; Clinical , Radiological and Microbiological Assesment
Brief Title: Role of Bronchoscopy in Bronchiectasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Yassin Ibrahim, Principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Bronchoscopy in bronchiectasis
Record Dates: First submitted 2019-09-21; First posted 2019-12-23 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Bronchoscopy
MeSH Terms: interventions — Bronchoscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Patients with bronchiectasis
  Interventions: Procedure: Bronchoscopy

INTERVENTIONS:
Procedure: Bronchoscopy — Role of bronchoscopy in diagnosis of bronchiectasis

SUMMARY:
Role of bronchoscopy in diagnosis of bronchiectasis in to different types

DETAILED DESCRIPTION:
Bronchiectasis is defined as abnormal chronic dilatation of one or more bronchi. Patients have a structural abnormality of the bronchial wall that predisposes them to bacterial infection likely due to impaired mucus clearance. A self-perpetuating vicious cycle of chest infections and chronic lung inflammation can lead to further damage of the bronchial wall and spread of disease to normal areas of bystander lung.(1)( Wilson et al,1997).

A search for an underlying cause, which may be amenable to a targeted intervention to prevent ongoing damage, is essential but often fruitless, and the focus of therapy rapidly turns to empiric treatments to prevent infective exacerbations and retard disease progression. (2) ( Martinez-Garcia, et al,2005 ) The British Thoracic Society bronchiectasis management guidelines provide an in-depth summary of the available literature and are an excellent tool for guiding treatment decision making. However, they do not provide guidance on which patients are most likely to benefit from specific interventions. (3) (Pasteur et al, 2010).

Disease severity in bronchiectasis is hard to define. Radiological severity grading scores exist; however, there is often a disconnect between radiological severity, symptom burden and disease progression (4) (Eshed et al, 2007).

In 2014, competing bronchiectasis severity scores were published (FACED and the Bronchiectasis Severity Index (BSI). In each of these, a combination of patient demographics, symptom scores, comorbidities, and clinical, radiological and microbiological parameters were used to construct scoring systems, which, in the case of the BSI, predicted future mortality, and in the case of FACED, extended to prediction of future exacerbation frequency, hospitalisation and quality of life. (5, 6) (Chalmers et al, 2014; Martinez-Garcia et al, 2014).

These severity scores have utility in identifying an individual's risk of disease progression to a predefined outcome and aid in subclassifying this heterogeneous group of patients in a manner that may pave the way to future mechanistic studies, which explain how these different disease phenotypes arise and inform the development of targeted therapeutics. (7) (Aliberti et al, 2007).

ELIGIBILITY:
Inclusion Criteria:

* patients more than 18 years
* Patients less than 70 years
* Patients with bronchiectasis

Exclusion Criteria:

* patients with bronchial asthma or chronic obstructive pulmonary disease
* patients with pneumonia
* patients with T.B

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of bronchiectatic patients with pseudomonal infection | One week
  Bronchoscopy will be done to all patients and bronchoalveolar lavage will be taken